CLINICAL TRIAL: NCT04479787
Title: Dorsal Spinal Cord Stimulation vs Medical Management for the Treatment of Low Back Pain (DISTINCT)
Brief Title: Spinal Cord Stimulation vs. Medical Management for Low Back Pain (DISTINCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10343
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low-Back Pain; Refractory Pain; Neuropathic Pain
Keywords: Chronic Low Back Pain; Spinal Cord Stimulation
MeSH Terms: conditions — Pain, Intractable; Neuralgia | interventions — Spinal Cord Stimulation; Physical Therapy Modalities; Dosage Forms; Injections; Acupuncture Therapy; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Spinal Cord Stimulation (SCS) (Active Comparator): An SCS Trial period followed by SCS Implantation with the Abbott Proclaim XR Implantable Pulse Generator
  Interventions: Device: Spinal Cord Stimulation
- Conventional Medical Management (CMM) (Active Comparator): CMM consists of an array of therapies including, but not limited to structured physical therapy, medications, injections, and complementary and alternative medicine (e.g. acupuncture, massage therapy)
  Interventions: Other: Conventional Medical Management

INTERVENTIONS:
Device: Spinal Cord Stimulation — Utilization of BURSTDR stimulation
  Other Names: Proclaim XR IPG
  Arms: Spinal Cord Stimulation (SCS)
Other: Conventional Medical Management — Assessing type of CMM, location and frequency.
  Other Names: Physical Therapy, Medications, Injections, Acupuncture, Massage Therapy, Etc.
  Arms: Conventional Medical Management (CMM)

SUMMARY:
The objective of this study is to evaluate the efficacy of BurstDR dorsal column stimulation, compared with conventional medical management, in improving pain and back-related physical function in subjects suffering with chronic, refractory axial low back pain with a neuropathic component, who have not had lumbar spine surgery and for whom surgery is not an option.

DETAILED DESCRIPTION:
A prospective, multi-center, randomized, controlled clinical study with an optional crossover component. The study is designed to evaluate the efficacy of BurstDR SCS in the treatment of chronic axial low back pain with a neuropathic component, compared to conventional medical management (CMM).

Subjects will be followed in-clinic at 1,3, 6, 9, 12, 18 and 24 months and via phone call or optional clinic visit at 15- and 21-months. The primary endpoint will be assessed at the 6-month follow-up visit. Upon completion of the 6-month follow-up visit, subjects who are dissatisfied with therapy and receiving inadequate improvement with their treatment assignment will be allowed to cross-over to the other treatment arm, if desired.

The study will enroll up to 270 patients at up to 30 sites. Subjects will be randomized in a 3:2 fashion to yield approximately 200 evaluable subjects for the primary endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be willing and able to provide written informed consent prior to any clinical investigation-related procedure.
2. Age ≥ 18 years
3. Patient has chronic (at least 6 months), refractory axial low back pain with a neuropathic component and is not a candidate for spine surgery
4. Patient has back pain for ≥ 6 months inadequately responsive to supervised conservative care
5. Patient has not had spine surgery for back or leg pain
6. Patient is a candidate for spinal cord stimulation
7. Low back pain ≥ 6 on Numerical Rating Scale
8. Oswestry Disability Index score of ≥ 30%
9. Willing and able to comply with the instructions for use, operate the study device, and comply with this Clinical Investigation Plan

Exclusion Criteria:

1. Pathology seen on imaging tests obtained within the past 12 months that is clearly identified and is likely the cause of the CLBP, that can be addressed with surgery.
2. Primary complaint of leg pain, or leg pain is greater than back pain
3. Back pain is due to any of the following:

   * spinal instability defined as > 2 mm translation on radiographic imaging
   * visceral causes (e.g., endometriosis or fibroids)
   * vascular causes (e.g., aortic aneurysm)
   * spinal infection (e.g., osteomyelitis)
   * inflammation or damage to the spinal cord (e.g. arachnoiditis or syringomyelia)
   * tumor or spinal metastases
4. Has widespread pain (e.g. fibromyalgia) or pain in other area(s), not intended to be treated in this study (e.g. neck pain, shoulder pain)
5. Patient has seronegative spondyloarthropathy (e.g. rheumatoid, lupus, psoriatic)
6. Neurological deficit (e.g. foot drop)
7. Prior lumbar spine surgery or sacroiliac joint fusion
8. Patient has used a morphine equivalent daily dose of more than 50 MME in the last 30 days
9. Patient is bed bound
10. Patients with regular intake of systemic steroids (except inhaled steroids used to treat asthma)
11. Imaging (MRI, CT, X-ray) findings within the last 12 months that contraindicates lead placement
12. Known allergic reaction to implanted materials
13. Severe scoliotic deformity (>11 degrees in thoracic or lumbar spine)
14. Patient has a history of, or existing intrathecal drug pump
15. Patient has previous experience with neuromodulation devices, including a failed trial
16. BMI > 40
17. Patient is enrolled, or intends to participate, in another clinical drug and/or device study or registry that may interfere with the results of this study, as determined by Abbott personnel
18. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results.
19. Failed psychological evaluation
20. Suspicion or evidence of untreated mental illness, or substance abuse
21. Patient demonstrated 2 or more Waddell's signs of nonorganic behavior
22. Patient is in current litigation for back pain/injury, or is currently receiving worker's compensation
23. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.

    * Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to enrollment/baseline visit per site standard test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yue, MD, Principal Investigator
Locations (30):
- United States (30):
  - Barrow Brain & Spine, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Spanish Hills Interventional Pain Specialists, Camarillo, California
  - Coastal Pain & Spinal Diagnostics Medical Group, Carlsbad, California
  - Napa Valley Orthopedic Medical Group, Napa, California
  - Connecticut Orthopedic Specialists, Hamden, Connecticut
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - The Orthopedic Institute, Gainesville, Florida
  - Anesthesia Pain Care Consultants, Tamarac, Florida
  - Axis Spine Center, Coeur d'Alene, Idaho
  - Chicago Anesthesia Associates, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Goodman Campbell Brain & Spine, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis Pain Consultants, Chesterfield, Missouri
  - Advanced Pain Care, Henderson, Nevada
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Albany Medical Center, Albany, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Spinal Diagnostics, Tualatin, Oregon
  - Center for Interventional Pain & Spine, Exton, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Carolina Orthopedics and Neurosurgical Associates, Spartanburg, South Carolina
  - Burkhart Research Institute for Orthopaedics, San Antonio, Texas
  - The Spine & Nerve Center of St Francis Hospital, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deer T, Gilligan C, Falowski S, Desai M, Pilitsis J, Jameson J, Moeschler S, Heros R, Tavel E, Christopher A, Patterson D, Wahezi S, Weisbein J, Antony A, Funk R, Ibrahim M, Lim C, Wilson D, Fishell M, Scarfo K, Dickerson D, Braun E, Buchanan P, Levy RM, Miller N, Duncan J, Xu J, Candido K, Kreiner S, Fahey ME, Yue J. Treatment of Refractory Low Back Pain Using Passive Recharge Burst in Patients Without Options for Corrective Surgery: Findings and Results From the DISTINCT Study, a Prospective Randomized Multicenter Controlled Trial. Neuromodulation. 2023 Oct;26(7):1387-1399. doi: 10.1016/j.neurom.2023.07.009. Epub 2023 Aug 28. PMID 37642628
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient enrolled in July 2020 was screen failed. Post that, the study enrolled the first subject in September, 2020. In total, 269 subjects were randomized at 30 investigational sites: 162 to SCS and 107 to CMM.
Period: Through 6 Months
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Started | 162 | 107
The Number of Subjects Implanted | 115 | 103
Cross Over to Alternate Arm | 0 | 70
Completed | 104 | 85
Not Completed | 58 | 22
Not completed — Withdrawal by Subject | 16 | 14
Not completed — Unsuccessful Trial | 17 | 0
Not completed — Subject Participation Terminated By Investigator | 12 | 3
Not completed — IPG/Lead(s) Explanted But Not Replaced | 2 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 3 | 0
Not completed — Inclusion/Exclusion | 2 | 1
Not completed — Subject Became Pregnant | 1 | 1
Not completed — Patient Diagnosed With Oral Cancer, Needs To Undergo Radiation And Chemo | 0 | 1
Not completed — Withdrawn At Sponsor's Request | 1 | 0
Not completed — Subject Failed To Comply With The Protocol Requirements | 1 | 0
Period: After 6 Months
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Started | 104 | 85
Completed | 94 | 54
Not Completed | 10 | 31
Not completed — Withdrawal by Subject | 3 | 13
Not completed — Unsuccessful Trial | 0 | 7
Not completed — IPG/Lead(s) Explanted But Not Replaced | 2 | 4
Not completed — Subject Participation Terminated By Investigator | 2 | 2
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Patient Was Withdrawn Due To Study Timelines | 0 | 1
Not completed — Patient's Health Significantly Declined | 0 | 1
Not completed — Subject Had Back Surgery On March 1st | 0 | 1
Not completed — Subject Failed To Comply With The Protocol Requirements | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants includes only the implanted patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM) | Total
Number analyzed (Participants) | 115 | 103 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number of participants analyzed includes only the implanted patients who completed the demographics questionnaire including age, sex, and race.
  years | 58.1 (13.0) | 59.1 (12.4) | 58.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes only the implanted patients who completed the demographics questionnaire including age, sex, and race.
  Participants
    Female | 69 | 52 | 121
    Male | 46 | 51 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes only the implanted patients who completed the demographics questionnaire including age, sex, and race.
  Participants
    White | 96 | 84 | 180
    Black or African American | 7 | 3 | 10
    Asian | 0 | 7 | 7
    American Indian or Alaska Native | 1 | 2 | 3
    Declined or Unable to Disclose Due to Local Regulation | 10 | 6 | 16
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    More than one race (One subject having both White and Asian race) | 0 | 1 | 1
Pain Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: scores on a scale] — Population: The number of participants analyzed includes only the implanted patients who completed the questionnaire for Pain Numeric Rating Scale.
  scores on a scale
    Lower Back | 7.7 (1.2) | 7.9 (1.1) | 7.8 (1.2)
    Right Leg: number analyzed (Participants) | 97 | 95 | 192
    Right Leg | 2.7 (2.6) | 3.1 (2.8) | 3.0 (2.7)
    Left Leg: number analyzed (Participants) | 100 | 94 | 194
    Left Leg | 2.8 (2.7) | 3.0 (2.8) | 3.0 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Responders Between Both Groups
Description: Improvement in pain, defined as percentage of patients who report a ≥ 50% decrease on Numeric Rating Scale (NRS).
Time Frame: 6 Months
Population: Percentage of patients who reported a 50% decrease in NRS pain score.
Measure: Number; unit: participants
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 119 | 81
participants | 87 | 5
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sided Z-Test

2. Secondary Outcome: Measure of Composite Responder Rate
Description: Composite Responder rate describes percentage of patients who responded on NRS OR ODI improvements (percentage of patients who report at least ≥13 change on ODI from baseline OR a ≥ 50% decrease in NRS from baseline).
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: participants
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 102 | 81
participants | 93 | 13
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sided Z-Test

3. Secondary Outcome: Numerical Rating Scale (NRS) Relative Change From Baseline to 6 Months
Description: The numeric rating scale (NRS) is a verbal or written determination of a pain level on a scale from 0 to 10, in which 0 represents no pain and 10 represents excruciating pain (the worst pain imaginable). Lower scores indicate pain reduction. The data is expressed as relative change (%).
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 102 | 81
percent change | 69.7 (24.9) | 5.6 (21.3)
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sample t-test

4. Secondary Outcome: Oswestry Disability Index (ODI) Change From Baseline to 6 Months
Description: The Oswestry Disability Index questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. An interpretation of 0% to 20% means minimal disability;21% to 40% means moderate disability; 41% to 60% means severe disability; 61% to 80% means crippled; and 81%-100% means bed-bound patients. Lower scores indicate less disability.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 98 | 81
units on a scale | 29.4 (18.8) | 0.7 (13.0)
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sample t-test

5. Secondary Outcome: Pain Catastrophizing Scale (PCS) Responder Rate
Description: The Pain Catastrophizing Scale questionnaire is a three part question that measures three pain domains:
  1. Rumination (e.g. "I can´t stop thinking about how much it hurts")
  2. Magnification (e.g. "I´m afraid that something serious might happen")
  3. Helplessness (e.g. "There is nothing I can do to reduce the intensity of my pain"). The Pain Catastrophizing Scale questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The questionnaire includes 13 statements describing different thoughts and feelings that may be associated with pain. Using the scale 0-4 (0- not at all; 1- to a slight degree; 2- to a moderate degree; 3- to a great degree; and 4- all the time), the patients are expected to indicate the degree to which they have these thoughts and feelings when they're experiencing pain. Lower scores indicate less catastrophizing thoughts.
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: participants
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 102 | 81
participants | 90 | 19
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sided Z-Test

6. Secondary Outcome: Patient Global Impression of Change (PGIC) Responder Rate
Description: PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." The percentage of patients who reported "very much improved," or "much improved," are presented.
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis. PGIC- % of patients who reported "very much improved," or "much improved."
Measure: Number; unit: participants
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 102 | 81
participants | 77 | 2
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sided Z-Test

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Pain Interference Relative Change From Baseline to 6 Months
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the pain interference domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome). Pain Interferences: Normal: <55; Mild: 55 - 60; Moderate: 60 -70; and Severe: >70.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 102 | 81
scores on a scale | 17.9 (11.3) | 0.9 (9.3)
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sample t-test

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Physical Function Relative Change From Baseline to 6 Months
Description: The PROMIS-29 physical function sub-scale includes 4 questions. The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the physical function domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., better outcome). Physical function- Normal: >45; Mild: 40 - 45; Moderate: 30 - 40; and Severe: >30.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
Number analyzed (Participants) | 102 | 81
scores on a scale | 27.8 (24.4) | 1.4 (13.6)
Statistical Analysis 1: Comparison: Spinal Cord Stimulation (SCS) vs Conventional Medical Management (CMM); Test type: Other; p < 0.0001, Two-sample t-test

ADVERSE EVENTS:
Time Frame: 6 months
Description: The CMM arm did not report any adverse event. The adverse events provided are all reported for the SCS arm.
Arm/Group | Spinal Cord Stimulation (SCS) | Conventional Medical Management (CMM)
All-Cause Mortality (participants affected / at risk) | 5/162 | 0/107
Serious Adverse Events (participants affected / at risk) | 7/162 | 0/107
Other Adverse Events (participants affected / at risk) | 17/162 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Cord Stimulation (SCS) (N=162) | Conventional Medical Management (CMM) (N=107)
Infection (Infections and infestations) | 2 | 0
Digoxin Toxicity (Injury, poisoning and procedural complications) | 1 | 0
Bladder Rupture (Renal and urinary disorders) | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Numbness Below The Level Of Implant (Surgical and medical procedures) | 1 | 0
Post Surgical Pain (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Cord Stimulation (SCS) (N=162) | Conventional Medical Management (CMM) (N=107)
Infection (Infections and infestations) | 3 | 0
Sleeping Issues And Weird Dreams (General disorders) | 1 | 0
Cerebrospinal Fluid (CSF) Leakage (Nervous system disorders) | 1 | 0
Changes In Stimulation Or Reduced Pain Relief Due To Lead Migration (Product Issues) | 4 | 0
Damage To The IPG Or Leads (General disorders) | 1 | 0
Dermatitis And Desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Implant Migration (General disorders) | 1 | 0
Movement Or Vibration Of The IPG Or Leads (General disorders) | 1 | 0
Persistent Pain At The IPG Site (General disorders) | 3 | 0
Skin Reaction (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT04479787/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT04479787/SAP_002.pdf